CLINICAL TRIAL: NCT00310440
Title: An Assessment of P-15 Bone Putty in Anterior Cervical Fusion With Instrumentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CeraPedics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1003
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Intervertebral Disk Degeneration
Keywords: Degenerative disc disease; P-15 Bone Putty; Bone graft; Cervical discectomy; Cervical spine
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone graft substitute (Experimental): Subjects will receive anterior cervical discectomy with fusion and instrumentation (anterior plate). Structural allograft ring will be used. The cavity of the ring will be filled with P-15 synthetic osteoconductive bone substitute (investigational device).
  Interventions: Device: P-15 Synthetic osteoconductive bone substitute
- Autologous Bone (Active Comparator): Subjects will receive anterior cervical discectomy with fusion and instrumentation (anterior plate). Structural allograft ring will be used. The cavity of the ring will be filled with local autologous bone.
  Interventions: Other: Autologous bone

INTERVENTIONS:
Device: P-15 Synthetic osteoconductive bone substitute — Safety and efficacy of synthetic bone substitute used for fusion in spinal surgery
  Other Names: i-Factor
  Arms: Bone graft substitute
Other: Autologous bone — Local autologous bone will be harvested, milled and placed into the cavity of the structural allograft ring
  Arms: Autologous Bone

SUMMARY:
The aim of this trial is to evaluate if P-15 bone putty (investigational device) is not inferior in effectiveness and safety to local autologous bone (control device) when applied in instrumented anterior cervical discectomy and fusion (ACDF) with use of a structural allograft ring in patients with degenerative cervical disc disease..

DETAILED DESCRIPTION:
Anterior Cervical Discectomy and Fusion (ACDF) is a common surgical treatment option for symptomatic degenerative cervical disk disease in patients who fail conservative treatment. i-FACTOR bone graft is a unique anorganic bone mineral (ABM) and small peptide, P-15™. P-15 is a synthetic fifteen amino acid polypeptide that mimics the cell-binding domain of Type I human collagen and is responsible for osteogenic cell attachment via alpha2-beta1 integrins.

This is randomized, controlled, multi-center, prospective FDA IDE study conducted to assess the safety and effectiveness of i-FACTOR bone graft (Cerapedics, Inc. Westminster, CO) in patients treated with single level ACDF. Patients received i-FACTOR bone graft or local autologous bone inside a structural allograft.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Radiographically determined discogenic origin to include at least one of the following characteristics: degenerated/dark disc on MRI, decreased disc height compared to adjacent levels on radiographic film, CT, or MRI and disc herniation on CT or MRI
* Radicular symptoms by history and physical exam to include at least the following characteristics: Arm/shoulder pain, decreased flexes, decreased strength and abnormal sensation
* Pain level arm/shoulder >4 on 0-10 VAS
* Pain level neck >4 on 0-10 VAS
* Neck disability Index >30
* Involved discs between C3 and C7
* Undergoing anterior cervical fusion at a single level
* Failed to gain adequate relief from non-operative treatment
* Able and willing to give consent to participate in study
* Understand and read English at elementary level

Exclusion Criteria:

Systemic infection such as AIDS, HIV, and active hepatitis; Significant metabolic disease that in the surgeon's opinion might compromise bone growth such as osteoporosis or osteomalacia; Taking medication for the prevention of osteoporosis; Circulatory, cardiac, or pulmonary problems that could cause excessive surgical risk; Active malignancy; Nondiscogenic source of symptoms (e.g., tumor, etc.); Multiple level symptomatic degenerative disc disease; Previous cervical fusion; Previous cervical decompression at the same level; Acute cervical trauma or instability (i.e., subluxation > 3 mm on flexion/extension radiographic film); Undergoing treatment for tumor or bony traumatic injury to the cervical spine; Rheumatoid disease of the cervical spine; Myelopathy; Pregnant or planning to become pregnant in the next 2 years; Posterior cervical spine procedure scheduled; More than one level to be operated; Has a history of substance abuse (recreational drugs, alcohol); Is a prisoner; Is currently involved in a study of another investigational product for similar purpose; Has a disease process that would preclude accurate evaluation (e.g., neuromuscular disease, significant psychiatric disease).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2006-01; Primary Completion 2014-05 (Actual); Study Completion 2019-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Janssen, MD / DO, Principal Investigator — Spine Education Research Institute
Locations (12):
- United States (10):
  - Department of Neurological Surgery UCSF Spine Center, San Francisco, California
  - Spine Education Research Institute, Thornton, Colorado
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Orthopaedics Northeast/Midwest Spine Group, Fort Wayne, Indiana
  - Indiana Spine Group, Indianapolis, Indiana
  - Indianapolis Neurosurgical Group, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - New England Neurosurgical Associates, LLC, Springfield, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - University of Utah Orthopaedic Center, Salt Lake City, Utah
- Canada (2):
  - Foothills Medical Center, Calgary, Alberta
  - Montreal Neurological Institute, Montreal, Quebec

REFERENCES:
- [Derived] Arnold PM, Vaccaro AR, Sasso RC, Goulet B, Fehlings MG, Heary RF, Janssen ME, Kopjar B. Six-Year Follow-up of a Randomized Controlled Trial of i-FACTOR Peptide-Enhanced Bone Graft Versus Local Autograft in Single-Level Anterior Cervical Discectomy and Fusion. Neurosurgery. 2023 Apr 1;92(4):725-733. doi: 10.1227/neu.0000000000002290. Epub 2022 Dec 23. PMID 36700705

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bone Graft Substitute | Autologous Bone
Started | 165 | 154
Completed | 139 | 141
Not Completed | 26 | 13
Not completed — Lost to Follow-up | 17 | 8
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Missed 12 Month Visit | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bone Graft Substitute | Autologous Bone | Total
Number analyzed (Participants) | 165 | 154 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (9.7) | 45.7 (9.4) | 46.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 97 | 192
  Male | 70 | 57 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 157 | 150 | 307
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 151 | 144 | 295
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 26 | 55
  United States | 136 | 128 | 264

OUTCOME MEASURES:

1. Primary Outcome: Radiologic Fusion
Description: Successful fusion was based on roentgenographic examination showing: evidence of bridging trabecular bone between the involved motion segments, translational motion <3mm, and angular motion <5 degrees. If there was a lack of evidence of fusion on 12 month plain x-ray examination, a CT-scan was performed and final determination of the fusion status was made using the CT reading. The criteria for fusion on CT scans were: trabecular bone formation patterns within the intervertebral disc space and bridging bone formation that crosses the interspace.
Time Frame: 12 months
Population: All participants that have radiological data at 12 months including imputed data.
Measure: Number; unit: participants
Arm/Group | Bone Graft Substitute | Autologous Bone
Number analyzed (Participants) | 145 | 141
participants
  Fused | 129 | 121
  No Evidence of Fusion | 16 | 20

2. Primary Outcome: Change in of the Overall Neck Disability Index (NDI) Score From Baseline.
Description: The NDI consists of ten items addressing functional activities (personal care, lifting, reading, work, driving, sleeping, recreational activities), pain intensity, concentration and headache. For each item, there are six potential responses, describing increasing degrees of disability (no disability = 0 to total disability = 5). An overall NDI score, out of 100, is calculated by adding up the scores for each item and multiplying by two. A higher NDI score indicates greater disability.
Time Frame: 12 months
Population: Per protocol (PP) subjects were included in this analysis. Six subjects that had major protocol deviations with the potential to impact the primary endpoint results were not included in the PP population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Bone Graft Substitute | Autologous Bone
Number analyzed (Participants) | 161 | 152
units on a scale | 28.75 [25.81 to 31.69] | 27.40 [24.35 to 30.45]

3. Primary Outcome: Neurologic Success
Description: The neurological endpoint is a binary variable. Neurologic success was assessed in the motor, sensory and reflex domains specific for the cervical spine as follows: maintenance or improvement of motor function in the elbow flexors (i.e. biceps muscle), elbow extensors (i.e. triceps muscle) and wrist extensors of both arms; maintenance or improvement of sensory function of both arms; maintenance or improvement of reflexes of both arms as measured at biceps tendon, triceps tendon and brachioradialis (supinator) reflex AND absence of Babinski reflex (if not present prior to surgery). Worsening of neurological status (neurological failure) was defined as a permanent decline in the subject's neurological status based on adjudication of accumulated neurological data by an independent blinded evaluator.
Time Frame: 12 months
Population: The total number of observed subjects.
Measure: Number; unit: participants
Arm/Group | Bone Graft Substitute | Autologous Bone
Number analyzed (Participants) | 143 | 143
participants
  Yes | 134 | 133
  No | 9 | 10

4. Primary Outcome: Complications
Description: Any AE within 12 months of surgery.
Time Frame: 12 months
Population: All enrolled subjects.
Measure: Number; unit: participants
Arm/Group | Bone Graft Substitute | Autologous Bone
Number analyzed (Participants) | 165 | 154
participants
  Yes | 138 | 127
  No | 27 | 27

5. Secondary Outcome: Mean Change in Pain at Neck Visual Analog Scale (VAS).
Description: The pain VAS is a continuous scale upon which the subject indicates their pain level ranging from "No pain at all" (0) to "Worst imaginable pain" (10). The change in pain is calculated by subtracting the 12 month score from the baseline score.
Time Frame: Baseline and 12 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Bone Graft Substitute | Autologous Bone
Number analyzed (Participants) | 161 | 152
cm | 4.45 [4.00 to 4.90] | 4.39 [3.96 to 4.82]

6. Secondary Outcome: Mean Change at Pain at Arm and Shoulder Visual Analog Scale (VAS).
Description: as for outcome 5
Time Frame: Baseline and 12 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Bone Graft Substitute | Autologous Bone
Number analyzed (Participants) | 161 | 152
cm | 4.89 [4.44 to 5.34] | 4.85 [4.40 to 5.30]

7. Secondary Outcome: Success Rates Measured by Aggregated Modified Odom's Criteria
Description: Subjects selected one of four categories: Excellent (Improvement Greater than or Equal to 80%, Deterioration Less than 10%), Good (Improvement Greater than or Equal to 70%, Deterioration Less than 15%), Fair (Improvement Greater than or Equal to 50%, Deterioration Less than 20%) or Poor (Improvement Less than 50%, Deterioration Greater than 20%).
Time Frame: 12 months
Population: Per protocol (PP) subjects that had data available at the 12 month visit were included in this analysis. Six subjects that had major protocol deviations with the potential to impact the primary endpoint results were not included in the PP population.
Measure: Number; unit: participants
Arm/Group | Bone Graft Substitute | Autologous Bone
Number analyzed (Participants) | 129 | 129
participants
  Excellent: Improvement GE 80% Deterioration LT 10% | 80 | 80
  Good: Improvement GE 70% Deterioration LT 15% | 25 | 25
  Fair: Improvement GE 50% Deterioration LT 20% | 16 | 15
  Poor: Improvement LT 50% Deterioration GT 20% | 8 | 9

8. Secondary Outcome: Mean Change in the Short Form 36 v2 (SF-36v2) Physical Composite Score (PCS).
Description: The SF-36 v2 (Medical Outcomes Trust, Boston, MA) is a multipurpose, patient-reported short-form health survey with 36 questions available in several languages. It yields two composite scores: one for physical health (Physical Composite Score - PCS) and one for mental health (Mental Composite Score - MCS) that are comprised of eight domains. The following domains make up the PCS: physical functioning, role-physical, bodily pain, general health. The PCS ranges from a score of 0 (lowest possible level of functioning) to a score of 100 (highest possible level of functioning).
Time Frame: Baseline and 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Bone Graft Substitute | Autologous Bone
Number analyzed (Participants) | 161 | 152
units on a scale | 10.02 [8.39 to 11.66] | 9.95 [8.25 to 11.65]

9. Secondary Outcome: Mean Change in the Short Form 36 v2 (SF-36v2) Mental Health Composite Score (MCS).
Description: The SF-36 v2 (Medical Outcomes Trust, Boston, MA) is a multipurpose, patient-reported short-form health survey with 36 questions available in several languages. It yields two composite scores: one for physical health (Physical Composite Score - PCS) and one for mental health (Mental Composite Score - MCS) that are comprised of eight domains. The following domains make up the MCS: vitality, social functioning, role-emotional, mental health. The MCS ranges from a score of 0 (lowest possible level of functioning) to a score of 100 (highest possible level of functioning).
Time Frame: Baseline and 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Bone Graft Substitute | Autologous Bone
Number analyzed (Participants) | 161 | 152
score on a scale | 8.33 [6.66 to 10.01] | 8.21 [6.48 to 9.95]

10. Secondary Outcome: Kyphosis
Description: Kyphosis is evaluated in degrees.
Time Frame: 12 months
Population: Per protocol (PP) subjects who had images available at 12 months were included in this analysis. Six subjects that had major protocol deviations with the potential to impact the primary endpoint results were not included in the PP population.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Bone Graft Substitute | Autologous Bone
Number analyzed (Participants) | 113 | 116
degrees | 3.0 (5.0) | 3.8 (4.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at all visits between baseline and 24 months.
Arm/Group | Bone Graft Substitute | Autologous Bone
Serious Adverse Events (participants affected / at risk) | 45/165 | 35/154
Other Adverse Events (participants affected / at risk) | 136/165 | 128/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Graft Substitute (N=165) | Autologous Bone (N=154)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 9 (10) | 8 (9)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 3 (4)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1)
Radiculitis cervical (Nervous system disorders) | 1 (1) | 0 (0)
Thoracic outlet syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1) | 3 (3)
Shoulder operation (Surgical and medical procedures) | 1 (1) | 2 (2)
Limb operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Arthroscopic surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Elbow operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrointestinal surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (2) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Nasal septal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Rotator cuff repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Uterine operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radial nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Implant site effusion (General disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Graft Substitute (N=165) | Autologous Bone (N=154)
Neck pain (Musculoskeletal and connective tissue disorders) | 67 (90) | 73 (100)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 (36) | 23 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (27) | 25 (28)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23 (26) | 21 (23)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 (15) | 22 (25)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 17 (20) | 18 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 10 (10)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 13 (15) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 8 (8)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 (5) | 11 (12)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 6 (9) | 10 (12)
Radiculopathy (Nervous system disorders) | 48 (75) | 55 (74)
Headache (Nervous system disorders) | 17 (18) | 23 (29)
Hypoaesthesia (Nervous system disorders) | 14 (16) | 20 (27)
Carpal tunnel syndrome (Nervous system disorders) | 12 (12) | 9 (11)
Paraesthesia (Nervous system disorders) | 7 (8) | 12 (14)
Dysphagia (Gastrointestinal disorders) | 31 (32) | 30 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less